CLINICAL TRIAL: NCT02007447
Title: Oxytocin in Adolescents With Autism Spectrum Disorders
Acronym: OXYASD
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Most of our patients had no willingness to participate in the survey
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Helena Paula Brentani, Helena Paula Brentani, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE 10922213.7.0000.0068
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Autism Spectrum Disorder
Keywords: autism, oxytocin, autism spectrum disorder, social skills.
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Social Skills | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OCYTOCINA - SPRAY NASAL (Active Comparator): OCYTOCINA - SPRAY NASAL - 24Ui twice per day for 8 weeks
  Interventions: Drug: OCYTOCINA - SPRAY NASAL
- Placebo (Placebo Comparator): Placebo - twice per day for 8 weeks
  Interventions: Drug: OCYTOCINA - SPRAY NASAL

INTERVENTIONS:
Drug: OCYTOCINA - SPRAY NASAL — The initial sample is divided into two groups (A and B): group A receive oxytocin intranasal for 8 weeks 24UI twice a day (3 applications per nostril 4UI 12/12 hours); group B will receive placebo for 8 weeks
  Other Names: SYNTOCINON - SPRAY NASAL; OXYTOCIN

SUMMARY:
This study is design to evaluate the influence of oxytocin in some aspects of Autism Spectrum Disorder (ASD), such as, repetitive and stereotyped behavior, social skills, quality of life and disruptive behaviors.

Null hypothesis: social skills, quality of life, disruptive behaviors and repetitive behaviors do not improve with the use of oxytocin. Experimental Hypothesis: social skills, quality of life, disruptive behaviors and repetitive and stereotyped behaviors improve with the use of oxytocin.

DETAILED DESCRIPTION:
Individuals with ASD have impaired social interaction, repetitive and disruptive behaviors. Oxytocin has been described to improve those skills and studies suggest that administration can reduce repetitive behaviors as well as enhance social interaction and communication deficits.

This study is design to evaluate the influence of oxytocin in some aspects of Autism Spectrum Disorder (ASD), such as, repetitive and stereotyped behavior, social skills, quality of life and disruptive behaviors.

Instruments:

1. Evaluation of social skills: Matson Evaluation of Social Skills (MESSY): consisting of 62 items divided into six factors that assess social skills such as appropriate social skills, assertiveness inadequate, impulsivity, self-confidence, jealousy withdraw, and other items that do not fit another classification.
2. Evaluation of repetitive behavior: Repetitive Behavior Scale (RBS): Consists of 43 items divided into six subscales: stereotyped behavior, self-harm behavior, compulsive behavior, ritualistic behavior, behavior monotonous and restricted behavior. This scale is able to measure the presence and severity of repetitive behaviors as common in individuals on the autism spectrum.
3. Evaluation disruptive behavior: Vineland, just the part that assess disruptive behavior
4. Multidimensional Student's Life Satisfaction Scale (MSLSS)

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 11 years 11 months and 17 years 11 months
* Autism spectrum disorder according to DSM V
* ADI > 10
* WISC > 70
* CARS > 30

Exclusion Criteria:

* Female
* presence of genetic and neurological syndromes
* changes in drugs or in any intervention during the study

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
SOCIAL SKILLS | 8 weeks
  Evaluation of social skills: Matson Evaluation of Social Skills (MESSY): consisting of 62 items divided into six factors that assess social skills such as appropriate social skills, assertiveness inadequate, impulsivity, self-confidence, jealousy withdraw, and other items that do not fit another classification.

SECONDARY OUTCOMES:
REPETITIVE BEHAVIOR | 8 WEEKS
  Evaluation of repetitive behavior: Repetitive Behavior Scale (RBS): Consists of 43 items divided into six subscales: stereotyped behavior, self-harm behavior, compulsive behavior, ritualistic behavior, behavior monotonous and restricted behavior. This scale is able to measure the presence and severity of repetitive behaviors as common in individuals on the autism spectrum.

OTHER OUTCOMES:
Evaluation disruptive behavior: Vineland, just the part that assess disruptive behavior | 8 WEEKS
  Evaluation disruptive behavior: Vineland, just the part that assess disruptive behavior
Multidimensional Student's Life Satisfaction Scale (MSLSS) | 8 WEEKS
  Multidimensional Student's Life Satisfaction Scale (MSLSS): SCALE OF QUALITY OF LIFE

CONTACTS AND LOCATIONS:
Overall Officials: Helena P. Brentani, PHD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Institute os Psychiatry, Clinical Hospital at São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tachibana M, Kagitani-Shimono K, Mohri I, Yamamoto T, Sanefuji W, Nakamura A, Oishi M, Kimura T, Onaka T, Ozono K, Taniike M. Long-term administration of intranasal oxytocin is a safe and promising therapy for early adolescent boys with autism spectrum disorders. J Child Adolesc Psychopharmacol. 2013 Mar;23(2):123-7. doi: 10.1089/cap.2012.0048. Epub 2013 Mar 12. PMID 23480321